CLINICAL TRIAL: NCT00515320
Title: Study Of Fluoxetine In Autism: A Randomised, Double-Blind, Placebo-Controlled, Parallel-Group 14-Week Study To Investigate The Effect Of Fluoxetine Orally Dissolving Tablet (ODT) On Repetitive Behaviors In Childhood And Adolescent Autistic Disorder.
Brief Title: Study of Fluoxetine in Autism
Acronym: SOFIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neuropharm (Industry)
Collaborators: Autism Speaks (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPL-2008-4-AUTUS-004
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Autistic Disorder
Keywords: Autism; children; adolescent; Fluoxetine; Autistic Disorder; Repetitive behavior; SSRI; Selective Serotonin Reuptake Inhibitor
MeSH Terms: conditions — Autistic Disorder | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine (Experimental)
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Once daily oral dispersible tablet 2mg 9mg or 18mg
  Other Names: NPL-2008
  Arms: Fluoxetine
Drug: Placebo — Oral dispersible tablet placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of fluoxetine orally dissolving tablets (ODT) on the repetitive behaviors core domain in children and adolescents with Autistic Disorder. The study will also investigate the effect of fluoxetine on the improvement of symptoms and the effects on daily living of the patient's family.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for autistic disorder, .
* CYBOCS-PDD score of at least 10 at screening.

Exclusion Criteria:

* Diagnosis of Asperger Syndrome or Pervasive Developmental Disorder Not Otherwise Specified, Rett Syndrome, Childhood Disintegrative Disorder.
* Patients planning to commence cognitive behaviour therapy during the period of the study or those who have begun cognitive behaviour therapy within 8 weeks prior to enrolment.
* Patients who are currently taking fluoxetine or who have previously taken it are not eligible for the study.

Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The percentage change from baseline to the endpoint visit for the CYBOCS-PDD score. | Throughout the study

SECONDARY OUTCOMES:
The time and dose related course of therapeutic effects | Throughout the study
The inter-relationship between these effects in the context of global clinical changes. | Throughout the study
The indirect effects on patient caregivers of the dose regime in these subjects compared to placebo during treatment. | Throughout the study
Safety measures will be physical examination, vital signs, EKG/ECG & clinical laboratory tests. | Throughout the study

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Southwest Autism Research and Resource Centre, Phoenix, Arizona
  - University of California Davis, Sacramento, California
  - University of Florida, Department of Psychiatry, Gainesville, Florida
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - University of Illinois, Chicago, Illinois
  - AMR-Baber Research Inc., Naperville, Illinois
  - Harvard Medical School, Medford, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - CRCNJ, Voorhees Township, New Jersey
  - Long Island Jewish Hospital, Bethpage, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Western Psychiatric Institute and Clinic/ Merck Child Outpatient Clinic, Pittsburgh, Pennsylvania
  - Red Oak Psychiatry Associates, Houston, Texas
  - Seattle Children's Hosptial University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Herscu P, Handen BL, Arnold LE, Snape MF, Bregman JD, Ginsberg L, Hendren R, Kolevzon A, Melmed R, Mintz M, Minshew N, Sikich L, Attalla A, King B, Owley T, Childress A, Chugani H, Frazier J, Cartwright C, Murphy T; Autism Speaks Autism Clinical Trials Network. The SOFIA Study: Negative Multi-center Study of Low Dose Fluoxetine on Repetitive Behaviors in Children and Adolescents with Autistic Disorder. J Autism Dev Disord. 2020 Sep;50(9):3233-3244. doi: 10.1007/s10803-019-04120-y. PMID 31267292
- See also: www.autismspeaks.org — http://www.autismspeaks.org